CLINICAL TRIAL: NCT00546988
Title: Multizentrische Therapiestudie Des Multiplen Myeloms DSMM V Therapieoptimierungs-Studie Der Deutschen Studiengruppe Multiples Myelom für Patienten Bis 60 Jahre im Stadium II/III
Brief Title: Multi Centre Trial of DSMM for Newly Diagnosed Multiple Myeloma up to 60 Years
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Wuerzburg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSMM V
Record Dates: First submitted 2007-10-17; First posted 2007-10-19 (Estimated); Last update posted 2007-10-19 (Estimated); Status verified 2007-10

CONDITIONS: Multiple Myeloma
Keywords: primary treatment; allogeneic stem-cell transplantation; high-dose therapy; cytogenetics
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Standard risk IFN (No Intervention): Administration of interferon alpha as a maintenance treatment following autologous stem cell transplantation
- Standard risk PEGIFN (No Intervention): Maintenance treatment with pegylated interferon following autologous stem cell transplantation
- High risk allo (Experimental): Allogeneic stem cell transplantation from an HLA identical related or unrelated donor
  Interventions: Biological: allogeneic stem cell transplant
- High risk auto (No Intervention): Second cycle of high-dose melphalan in subjects without an HLA-identical donor

INTERVENTIONS:
Biological: allogeneic stem cell transplant
  Arms: High risk allo

SUMMARY:
The study is evaluating whether risk-stratification by the means of a chromosomal aberration provides a tool to discriminate between standard and high risk. Risk-adapted therapy is based on allogeneic stem-cell transplantation for high-risk subjects instead of a second autograft in patients with deletion of chromosome 13 who have an HLA-identical stem cell donor available.

DETAILED DESCRIPTION:
The DSMM V protocol is to compare a consolidation treatment for standard-risk patients not displaying del(13) at initial diagnosis following two cycles of high-dose melphalan 200 mg/m² each supported by autologous stem cell retransfusion with interferon versus PEG-interferon. Patients with del(13) are screened for availability of a fully HLA-matched related or unrelated donor. If patient's informed consent is obtained additionally, he is scheduled to undergo an allogeneic SCT following the first cycle of high-dose melphalan. All other subjects are to proceed to a second course of high-dose melphalan similar to the standard-risk group. Initial cytoreduction is foreseen with four cycles of anthracycline-dexamethasone combination followed by combination therapy with ifosfamide/epirubicine/etoposide for stem-cell collection.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of multiple myeloma
* Salmon-and-Durie stage II or III
* Less than or equal to 60 years
* Signed informed consent

Exclusion Criteria:

* Relevant comorbidities
* Unable to adhere to study protocol
* Pregnancy
* Not received subject's informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2001-10; Study Completion 2008-01 (Estimated)

PRIMARY OUTCOMES:
Response rate after high-dose therapy | one year

SECONDARY OUTCOMES:
Response rate and treatment-related mortality after allogeneic transplantation | one year

CONTACTS AND LOCATIONS:
Overall Officials: Hermann Einsele, M.D., Principal Investigator — Wuerzburg University Hospital, Dept. of Hematology and Oncology
Locations (29):
- Austria (2):
  - Medizinische Univ.-Klinik Graz, Graz
  - Klin. Abt. für Onkologie, AKH Wien, Vienna
- Germany (27):
  - Staedtisches Klinikum, Augsburg
  - Dept. of Hematology/Oncology, Charité Berlin, Berlin
  - Charité University Medicine, Berlin
  - University Hospital, Erlangen
  - Krankenhaus Nordwest, Frankfurt
  - Freiburg University Hospital, Freiburg im Breisgau
  - Georg August University Hospital, Göttingen
  - Ernst-Moritz Arndt University Hospital, Greifswald
  - Martin-Luther University Hospital, Halle
  - University Hospital Eppendorf, Hamburg
  - Hannover Medical School, Hanover
  - Saarland University Hospital, Homburg/Saar
  - Schleswig-Holstein University Hospital, Lübeck
  - Mainz University Hospital, Mainz
  - Dept. of Internal Medicine, Ludwig-Maximilian-University Munich, Munich
  - Klinikum rechts der Isar, Munich
  - Dept. of Internal Medicine A, University Muenster, Münster
  - Nuremberg Central Hospital, Nuremberg
  - Oldenburg Hospital, Oldenburg
  - University Hospital, Regensburg
  - Katharinenhospital, Stuttgart
  - Diakonissenkrankenhaus, Stuttgart
  - Tubingen University Hospital, Tübingen
  - Dept. of Internal Medicine III, University of Ulm, Ulm
  - Ulm University Hospital, Ulm
  - Horst-Schmidt-Kliniken, Wiesbaden
  - Dept. of Internal Medicine II, University of Wuerzburg, Würzburg

REFERENCES:
- See also: Site of the German association of the leading research groups in lymphoid malignancies — http://www.lymphome.de